CLINICAL TRIAL: NCT07118514
Title: Effects of a Resistance Training Program on Immunological, Psychological, and Functional Indicators in People With Multiple Sclerosis: A Randomized Clinical Trial
Brief Title: Effect of Resistance Training on Psychophysiological Indicators in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of Maringá (Other)
Responsible Party: Principal Investigator, Cleverson José Bezerra Guedes, Principal Investigator, State University of Maringá
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 70726623.3.0000.0104
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; BDNF; Irisin; Anxiety; Depression; Exercise; Quality of life; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Anxiety Disorders; Depression; Motor Activity; Fatigue | interventions — Resistance Training; Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 2:1 ratio to either an intervention group (supervised progressive resistance training) or a control group (light stretching and relaxation activities). The intervention will last 12 weeks, with two sessions per week. All outcomes will be assessed at baseline and post-intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Participants in this group will undergo a 12-week supervised resistance training program, twice a week for approximately 50 minutes per session. Exercises are performed on fixed machines and based on 1-repetition maximum (1-RM) tests, with progressive loads from 50% to 65% of 1-RM. Training includes leg press, leg curl, knee extension, chest press, biceps and triceps curls, seated row, and lat pulldown
  Interventions: Behavioral: Progressive Resistance Training
- Control Group (Active Comparator): Participants in this group will engage in light stretching and relaxation sessions twice a week for 12 weeks. Each session lasts approximately 30-40 minutes and includes breathing exercises, stretching of major muscle groups, and guided relaxation.
  Interventions: Behavioral: Stretching and Relaxation Activities

INTERVENTIONS:
Behavioral: Progressive Resistance Training — A 12-week supervised resistance training program, performed twice weekly for 50 minutes per session. Exercises are based on 1-repetition maximum (1-RM) tests, using fixed machines and progressive loads (50-65% of 1-RM). Exercises include leg press, leg curl, knee extension, chest press, biceps/triceps curls, seated row, and lat pulldown.
  Other Names: Resistance training; Weight Training; Strength Training
  Arms: Exercise Group
Behavioral: Stretching and Relaxation Activities — A 12-week supervised program focused on flexibility and relaxation, performed twice weekly for approximately 50 minutes. Includes static stretching of major muscle groups and guided breathing exercises aimed at reducing muscle tension and promoting mental relaxation.
  Other Names: Static Muscle Stretching; Dynamic Stretching; Flexibility Protocols
  Arms: Control Group

SUMMARY:
This randomized controlled trial aims to investigate the effects of a supervised resistance training program on plasma levels of Brain-Derived Neurotrophic Factor (BDNF) and irisin in individuals diagnosed with multiple sclerosis (MS). The study will also examine secondary outcomes, including fatigue, quality of life, anxiety and depression symptoms, muscular strength, and functional capacity.

Participants will be randomly assigned to either an intervention or control group in a 2:1 allocation ratio. The intervention group will undergo a 12-week supervised resistance training program, while the control group will maintain their usual care without engaging in any structured exercise regimen. The trial will be non-blinded and involve assessments at baseline and after the 12-week intervention period.

Eligible participants must be adults (≥18 years), of any sex, with a confirmed diagnosis of MS by a neurologist, and currently undergoing disease-modifying therapy (DMT). Participants must not be engaged in any other structured physical exercise program, though symptom-management physiotherapy will be permitted. All participants should have sufficient mobility to complete the training sessions and assessments.

Exclusion criteria include the inability to perform the physical training or functional tests due to severe mobility restrictions, lack of standard pharmacological treatment for MS, or concurrent participation in other structured exercise programs.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the effects of a 20-week progressive resistance training program on psychophysiological parameters in individuals with multiple sclerosis (MS). The study compares a resistance-training intervention group with an active control group performing stretching and relaxation exercises, aiming to determine changes in hormonal, immunological, motor, and psychological outcomes.

MS is a chronic, immune-mediated demyelinating disease of the central nervous system, associated with neuroinflammation, neurodegeneration, and significant variability in clinical presentation. Common symptoms such as fatigue, depression, and motor impairment severely impact quality of life. Research suggests that exercise can promote neuroprotection, modulate inflammatory processes, and improve both physical and psychological well-being in this population.

The intervention is based on established exercise guidelines for mild to moderate MS and is adapted from protocols demonstrating safety and feasibility in this population. It seeks to investigate simultaneous effects on circulating biomarkers - including brain-derived neurotrophic factor (BDNF), irisin, vitamin D, cortisol, vascular endothelial growth factor (VEGF), nerve growth factor (NGF), neurotrophin-3 (NT-3), and neurotrophin-4 (NT-4) - alongside functional capacity, muscle strength, body composition, and validated measures of fatigue, quality of life, anxiety, depression, motivation, and habitual physical activity.

Assessments are conducted before and after the intervention period, with all laboratory analyses performed under standardized fasting and sample-processing conditions. Functional and psychological measures are obtained using validated instruments for the Brazilian population. Participants are monitored to ensure high adherence rates, with makeup sessions provided when possible.

This trial addresses a gap in the literature by jointly evaluating neurotrophic, hormonal, motor, and psychological responses to structured exercise in Brazilian individuals with MS, and by including an active control condition to account for the potential influence of social interaction and attention. The findings may inform future rehabilitation strategies and complement pharmacological management, contributing to improved patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Multiple Sclerosis (MS) according to the 2017 McDonald Criteria
* Expanded Disability Status Scale (EDSS) score between 1.0 and 6.0
* Age between 18 and 60 years
* Medical clearance to engage in physical exercise
* Ability to understand and provide written informed consent
* Stable pharmacological treatment for MS for at least 3 months prior to enrollment
* No MS relapses or corticosteroid use within 30 days before starting the intervention

Exclusion Criteria:

* Pregnancy or planning to become pregnant during the study period
* Severe musculoskeletal conditions contraindicating exercise
* Participation in another structured or systematic exercise program
* Visual, cognitive, or communication impairments that may hinder participation
* Use of orthopedic devices incompatible with the intervention protocols
* Any other condition that, in the opinion of the research team, may interfere with participation or compromise data integrity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Plasma levels of cortisol, brain-derived neurotrophic factor (BDNF), and irisin. | - Baseline - 12 weeks
  Change in plasma concentrations of cortisol, BDNF and irisin, measured using enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
Muscle Strength (Dynamic and Isokinetic) | - Baseline - 12 weeks
  Change in maximal strength of lower and upper limbs assessed by one-repetition maximum (1-RM) tests in selected exercises (e.g., leg press, chest press), and by isokinetic dynamometry of the knee extensors and flexors.
Functional Mobility | - Baseline - 12 weeks
  Change in mobility performance assessed by the Timed Up and Go (TUG) test.
Isokinetic Muscle Strength (Lower Limbs) | - Baseline -12 weeks
  Change in peak torque of knee extensors and flexors measured using isokinetic dynamometry at angular velocities of 60°/s and 180°/s.
Fatigue | - Baseline -12 weeks
  Change in fatigue perception measured by the Modified Fatigue Impact Scale (MFIS).
Anxiety and Depression | - Baseline -12 weeks
  Change in psychological symptoms assessed by the Hospital Anxiety and Depression Scale (HADS), including anxiety and depression subscales.
Health-Related Quality of Life | - Baseline - 12 weeks.
  Change in quality of life assessed by the Multiple Sclerosis Impact Scale (MSIS-29)
Optimism | - Baseline - 12 weeks.
  Change in dispositional optimism assessed by the Revised Life Orientation Test (LOT-R).
Perceived Barriers to Physical Activity | - Baseline .
  Change in perceived barriers assessed by the Barriers to Physical Activity Questionnaire (Petroski, 2000).
Physical Activity Level | - Baseline
  Change in habitual physical activity level assessed by the Baecke Habitual Physical Activity Questionnaire.
Motivation for Exercise | - Baseline
  Change in motivation for physical activity assessed by the Behavioral Regulation in Exercise Questionnaire-3 (BREQ-3).
Trait Anxiety Levels | - At baseline (before randomization) -12 weeks from the start of the intervention
  Assessment of trait anxiety levels using the State-Trait Anxiety Inventory - Trait subscale (STAI-T), validated for the Brazilian population. The instrument consists of 20 self-reported items rated on a Likert-type scale, with total scores ranging from 20 to 80 points; higher scores indicate greater trait anxiety.
  Time Frame:

CONTACTS AND LOCATIONS:
Locations (1):
- State University of Maringá, Maringá, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No